CLINICAL TRIAL: NCT06389409
Title: Observational Study on the Quality of Life and Functional/Oncological Outcome of Patients Undergoing Surgery for Testicular Removal and/or Removal of Retro-peritoneal Lymph Nodes
Brief Title: Study on the Quality of Life and Functional/Oncological Outcome of Testicular Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Salonia, Professor, IRCCS San Raffaele
Other Study IDs: Protocollo N.2009 Testicolo
Record Dates: First submitted 2024-02-20; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Testicular Cancer
Keywords: testicular cancer
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with testicular cancer: * subjects suffering from suspected neoplastic testicular pathology candidates for testicle removal surgery
  * patients suffering from neoplastic testicular pathology requiring removal of the retroperitoneal lymph nodes
  Interventions: Other: Observation of testicular cancer patients

INTERVENTIONS:
Other: Observation of testicular cancer patients — Collection of clinical data of all patients suffering from neoplastic testicular pathology undergoing surgery

SUMMARY:
The research aims to collect data in order to report the main problems related to the testicular cancer; To reach this aim, this study proposes to create a database of the testicular cancer condition.

From this perspective, the aim of this project is the improving of scientific knowledge of the disease and develop appropriate and effective procedures for the diagnosis and treatment of the patient.

DETAILED DESCRIPTION:
Testicular cancer constitutes 1% to 1.5% of male tumors, 5% of urological tumors. In the Western society to which we belong, the incidence is between 3 and 6 new cases per 100,000 inhabitants per year. In particular, this incidence has recorded continuous growth over the last thirty years. Different histologies of this disease are known, with a clear prevalence of germ cell tumors (90-95%).

From these general epidemiological coordinates it can be deduced that this pathology could affects a young segment of the population; It must be underlined that a pathology is peculiar due to the impact it has on the affected individual, who must be treated not only from an oncological point of view but also with regards to the sexual, reproductive and psychological-relational aspects. Such complexity requires a systematic and detailed approach to examine all aspects.

The creation of this database let to have a follow up above all an extension over time that is not present in the literature, especially towards the functional aspects of this condition.

The database will represent a resource for future research.

ELIGIBILITY:
Inclusion Criteria:

* subjects suffering from suspected neoplastic testicular pathology candidates for testicle removal surgery
* patients suffering from neoplastic testicular pathology requiring removal of the retroperitoneal lymph nodes
* subjects > 18 years old
* subjects with at least elementary education
* signature of informed consent

Exclusion Criteria:

* subjects < 18 years
* presence of mental or physical disability that may prevent the patient from satisfying the requirements of the protocol

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients suffering from neoplastic testicular pathology undergoing (or candidates for) surgery
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-08-24 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2040-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical data | Baseline
  Collection of clinical data
Adjuvant therapy | Baseline
  Which type of adjuvant therapy carried out (chemotherapy - radiotherapy - retroperitoneal lymphadenectomy)
lactate dehydrogenase | Follow up after 6 months from baseline
  Oncological follow-up through enzymatic value
Testicular objective examination | Baseline
  Number and size (via Prader orchidometer) of the testicles
Testicular objective examination - cysts | Baseline
  Evaluation presence of cysts
Testicular objective examination - nodules | Baseline
  Evaluation presence of nodules
Testicular objective examination - varicocele | Baseline
  Evaluation presence of varicocele
Testicular objective examination - hydrocele | Baseline
  Evaluation presence of hydrocele
α-feto protein | Follow up after 6 months from baseline
  Oncological follow-up through enzymatic value
β human Chorionic Gonadotropin | Follow up after 6 months from baseline
  Oncological follow-up through hormonal value
carcinoembryonic antigen | Follow up after 6 months from baseline
  Oncological follow-up through hormonal value

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Salonia, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No